CLINICAL TRIAL: NCT02919683
Title: Window Study of Nivolumab With or Without Ipilimumab in Squamous Cell Carcinoma of the Oral Cavity
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jonathan Schoenfeld, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-284
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab With Ipilimumab (Experimental): * Nivolumab to be delivered at a pre-determine dose for two weeks
  * Ipilimumab to be delivered at a pre-determine dose for one week
  * Blood Sample Collected
  * Standard of Care Surgery
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Procedure: Standard of Care Surgery
- Nivolumab (Experimental): * Nivolumab to be delivered at a pre-determine dose for two weeks
  * Blood Sample Collected
  * Standard of Care Surgery
  Interventions: Drug: Nivolumab; Procedure: Standard of Care Surgery

INTERVENTIONS:
Drug: Nivolumab
  Other Names: Opdivo
Drug: Ipilimumab
  Other Names: Yervoy
  Arms: Nivolumab With Ipilimumab
Procedure: Standard of Care Surgery

SUMMARY:
This research study is studying nivolumab, an investigational drug, in combination with ipilimumab, also an investigational drug, as a possible treatment for Squamous Cell Carcinoma of the oral cavity.

The following drugs are involved in this study:

* Nivolumab (Opdivo™)
* Ipilimumab (Yervoy™)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The purpose of this study is to evaluate effectiveness (how well the drug/s work) of Nivolumab or Nivolumab combined with Ipilimumab prior to standard of care surgery.

Nivolumab and Ipilimumab are types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells. Both nivolumab and Ipilimumab have been demonstrated to activate the immune system to attack cancer cells in laboratory studies and in patients with different types of cancers.

Nivolumab (Opdivo ™) has been approved by the US Food and Drug Administration (FDA) for the treatment of metastatic melanoma (a type of skin cancer), and specific types of previously treated advanced lung and kidney cancers. Ipilimumab (Yervoy™) is approved by the FDA for the treatment of metastatic melanoma.

Because Nivolumab and Ipilimumab help the immune system work in different ways, the combination of Nivolumab and Ipilimumab was tested in laboratory studies. The data from these studies suggested that giving the two drugs together could be of benefit to patients, and this was indeed found to be the case in patients with melanoma. The combination of Nivolumab and Ipilimumab is now FDA approved as treatment for patients with metastatic melanoma. However, the use of Nivolumab as well as Ipilimumab alone or in combination for the treatment of patients with head and neck cancer is not approved. Results from clinical trials investigating the safety and efficacy of Nivolumab and Ipilimumab in patients with head and neck cancer are not available at this time.

In the proposed study, either Nivolumab or the combination of Nivolumab and Ipilimumab is being tested is being tested prior to surgery to remove cancers of the oral cavity. By stimulating the immune system to attack cancer cells, these drugs may cause the cancer to decrease in size prior to surgery and prevent the cancer from coming back.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell carcinoma of the oral cavity. Clinical stage >=T2 (primary tumor greater than 2 cm in size) and/or evidence of regional nodal involvement by clinical exam or imaging
* Only patients 18 years and older are eligible. There is no upper age limit but the patients must be able to medically tolerate the regimen. Adverse event data are currently unavailable on the use immune checkpoint blockade for participants < 18 years of age, and thus children are excluded from this study
* ECOG performance status <=1
* Patients much be a surgical candidate (e.g. their disease must be considered resectable before any treatment and must have no serious medical contraindications that definitively preclude undergoing general anesthesia) Ability to understand and the willingness to sign a written informed consent document
* Women of childbearing potential (WOCBP) must agree to use appropriate method(s) of contraception (see Appendix B). WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. WOCBP is defined as any woman or adolescent who has begun menstruation and is not post- menopausal. A post-menopausal woman is defined as a woman who is over the age of 45 and has not had a menstrual period for at least 12 months
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab
* Men who are sexually active with WOCBP must agree to use any contraceptive method (see Appendix B) with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception)
* Participants must have normal organ and marrow function as defined below:

Laboratory parameters: WBC ≥ 2000/uL, Absolute neutrophil count (ANC) ≥ 1500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin (Hgb) ≥ 9 g/dL; Hgb-A1C ≤ 7.5%; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); Bilirubin ≤ 2.5 × ULN (≤ 4 × ULN for subjects with Gilbert's disease); Alkaline phosphatase ≤ 2.5 × ULN; Creatinine ≤ 1.5 × ULN

Exclusion Criteria:

* Pathologically proven, radiologic or clinical evidence of distant metastatic disease (this includes all disease below the clavicles, as well as disease metastatic to the bone, brain, or in the spinal canal)
* Any prior immunologic cancer therapy with systemic inhibitors of the PD-1 or CTLA-4 pathway
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; or if diagnosed and treated within the past 2 years for cervical cancer in situ or basal cell or squamous cell carcinoma of the skin
* Prior radiation to the head and neck region
* Prior chemotherapy within the last 2 years
* History of pneumonitis or interstitial lung disease
* Has evidence of active, noninfectious pneumonitis that required treatment with steroids.
* Active, suspected or prior documented autoimmune disease that has required systemic treatment in the last 2 years with immune modifying agents (e.g. replacement therapy such as thyroxine, insulin or physiologic corticosteroids is not an exclusion criteria). This does not include patients with vitiligo or type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* The subject is known to be positive for the human immunodeficiency virus (HIV), HepBsAg, or HCV RNA
* Lack of availability for follow up assessments
* Concurrent administration of other cancer specific therapy during the course of this study is not allowed
* Patients who require systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* The investigator's belief that the subject is medically unfit to receive nivolumab, and/or ipilimumab or unsuitable for any other reason
* Has received a live vaccine within 28 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2019-07 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Schoenfeld, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah H, Wang Y, Cheng SC, Gunasti L, Chen YH, Lako A, Guenette J, Rodig S, Jo VY, Uppaluri R, Haddad R, Schoenfeld JD, Jacene HA. Use of Fluoro-[18F]-Deoxy-2-D-Glucose Positron Emission Tomography/Computed Tomography to Predict Immunotherapy Treatment Response in Patients With Squamous Cell Oral Cavity Cancers. JAMA Otolaryngol Head Neck Surg. 2022 Mar 1;148(3):268-276. doi: 10.1001/jamaoto.2021.4052. PMID 35050348
- [Derived] Schoenfeld JD, Hanna GJ, Jo VY, Rawal B, Chen YH, Catalano PS, Lako A, Ciantra Z, Weirather JL, Criscitiello S, Luoma A, Chau N, Lorch J, Kass JI, Annino D, Goguen L, Desai A, Ross B, Shah HJ, Jacene HA, Margalit DN, Tishler RB, Wucherpfennig KW, Rodig SJ, Uppaluri R, Haddad RI. Neoadjuvant Nivolumab or Nivolumab Plus Ipilimumab in Untreated Oral Cavity Squamous Cell Carcinoma: A Phase 2 Open-Label Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1563-1570. doi: 10.1001/jamaoncol.2020.2955. PMID 32852531

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab With Ipilimumab: * Nivolumab to be delivered at a pre-determine dose for two weeks
  * Ipilimumab to be delivered at a pre-determine dose for one week
  * Blood Sample Collected
  * Standard of Care Surgery
  Nivolumab
  Ipilimumab
  Standard of Care Surgery
- Nivolumab: * Nivolumab to be delivered at a pre-determine dose for two weeks
  * Blood Sample Collected
  * Standard of Care Surgery
  Nivolumab
  Standard of Care Surgery
Period: Pre-Surgery Intervention
Arm/Group | Nivolumab With Ipilimumab | Nivolumab
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Post-Surgery Follow-Up
Arm/Group | Nivolumab With Ipilimumab | Nivolumab
Started | 15 | 15
Completed | 12 | 13
Not Completed | 3 | 2
Not completed — Death | 2 | 2
Not completed — Patient is still completing follow-ups | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab With Ipilimumab | Nivolumab | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Volumetric Response Rate to Treatment
Description: Response rate to window treatment with single agent nivolumab or nivolumab combined with ipilimumab is determined using bidirectional measurements (product of longest 2 diameters of lesions) of primary and nodal lesions to be removed at the time of surgery.
  Responders will have demonstrated any reduction in overall tumor volume as determined by the product of the longest perpendicular bidirectional tumor measurements.
Time Frame: At time of surgery
Population: Thirty patients were treated from 2016 to 2019. One patient was excluded from efficacy analyses as she was ineligible because of evidence of distant metastatic disease at baseline.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab With Ipilimumab | Nivolumab
Number analyzed (Participants) | 15 | 14
percentage of participants | 53 [34.2 to 71.8] | 50 [30.5 to 69.5]

2. Primary Outcome: Safety and Tolerability of Protocol Treatment
Description: Outcome measure includes number of participants with treatment-related adverse events as assessed by CTCAE v4.0, number of dose-limiting toxicities in safety run-ins following a 3 + 3 design, and delays to surgery.
Time Frame: At the time of surgery
Measure: Number; unit: instances
Arm/Group | Nivolumab With Ipilimumab | Nivolumab
Number analyzed (Participants) | 15 | 15
instances
  Delays to Surgery | 0 | 0
  Dose-Limiting Toxic Effects during Safety Run-In | 0 | 0
  Grade 3-4 Events At Least Possibly Related to Protocol Treatment | 5 | 2

3. Secondary Outcome: Percentage of Participants Demonstrating Objective Response Using RECIST Criteria
Description: Determining the radiologic response rate following the window treatment as determined by RECIST v1.1.
Time Frame: At time of surgery
Population: For this analysis, patients with no radiographically measurable lesions on imaging review were excluded. Thirty patients were treated from 2016 to 2019. One patient was excluded from efficacy analyses as she was ineligible because of evidence of distant metastatic disease at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab With Ipilimumab | Nivolumab
Number analyzed (Participants) | 13 | 14
percentage of participants | 38 | 13

4. Secondary Outcome: Percentage of Participants Demonstrating Pathological Response
Description: Pathologic response in the primary tumor was assessed using a quantitative grading scheme:
  pathologic tumor response [nonviable tumor] PTR0 = no or <10% response PTR1 = ≥10% PTR2 = ≥50%
Time Frame: At time of surgery
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab With Ipilimumab | Nivolumab
Number analyzed (Participants) | 15 | 14
percentage of participants
  PTR1 | 40 | 38
  PTR2 | 33 | 15

5. Secondary Outcome: Participant One Year Progression-Free Survival Percentage
Description: Progression-free survival is defined as the time between first study treatment and either recurrent disease or death. Recurrent disease includes a local failure, regional failure, or distant metastasis.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: All participants enrolled in both trial cohorts.
Arm/Group | All Participants
Number analyzed (Participants) | 29
percentage of participants | 85 [72.4 to 99.7]

6. Secondary Outcome: Participant Overall Survival Percentage
Description: Overall survival is defined as the time between first study treatment and death.
Time Frame: Data Cutoff (14.2 Months Median Follow Up)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 29
percentage of participants | 89 [78.3 to 100]

ADVERSE EVENTS:
Time Frame: All adverse events experienced by participants were collected from the time of the first dose of study treatment, through the study and until the final study visit 1 year after enrollment.
Description: The descriptions and grading scales found in the CTEP Active Version of the NCI Common Terminology Criteria for Adverse Events (CTCAE version 4.0) were utilized for AE reporting.
Arm/Group | Nivolumab With Ipilimumab | Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/15 | 2/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 3/15
Other Adverse Events (participants affected / at risk) | 12/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab With Ipilimumab (N=15) | Nivolumab (N=15)
Thromboembolic event (Vascular disorders) | 0 | 1
Right knee effusion and fever (Musculoskeletal and connective tissue disorders) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Wound complication - flap thrombosis and failure (Surgical and medical procedures) | 1 | 0
Stroke (Vascular disorders) | 1 | 0
hyperglycemia and diabetic ketoacidosis (Endocrine disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab With Ipilimumab (N=15) | Nivolumab (N=15)
Dysphagia (Gastrointestinal disorders) | 1 | 3
Oral pain (General disorders) | 3 | 5
Fatigue (General disorders) | 1 | 4
Hyperthyroidism (Endocrine disorders) | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 0
Osteonecrosis of the jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dental caries (General disorders) | 1 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pruitus (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Edema (General disorders) | 3 | 1
Dry mouth (General disorders) | 1 | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Autoimmune disorder (Immune system disorders) | 1 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Mucositis (Gastrointestinal disorders) | 2 | 1
Paresthesia (General disorders) | 0 | 2
Lymph node pain (General disorders) | 1 | 0
Fever (General disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Muscle/Joint Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Delayed wound healing (General disorders) | 0 | 1
Anorexia (General disorders) | 1 | 0
Lymphedema (General disorders) | 1 | 0
Oral ulcer (Gastrointestinal disorders) | 0 | 1
Glucose intolerance (General disorders) | 0 | 1
Infusion-related reaction (General disorders) | 1 | 0
Allergic Reaction (Immune system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT02919683/Prot_SAP_000.pdf